CLINICAL TRIAL: NCT02109393
Title: Rehabilitation in Patients With Progressive Supranuclear Palsy: Effectiveness of Two Intensive Protocols
Brief Title: Rehabilitation in Patients With Progressive Supranuclear Palsy
Acronym: PSP-MIRTLoko
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSP-MIRTLoko; PSP MIRT-Loko 001 (Other: Ospedale Generale di Zona "Moriggia-Pelascini")
Record Dates: First submitted 2014-03-25; First posted 2014-04-09 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-11

CONDITIONS: Progressive Supranuclear Palsy
Keywords: Rehabilitation; Robot-assisted walking training; Treadmill; Lokomat
MeSH Terms: conditions — Supranuclear Palsy, Progressive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MIRT group (Experimental): This group underwent a 4-weeks MIRT exploiting the use of a treadmill-plus (treadmill associated with visual cues and auditory feedbacks).
  Inclusion criteria: a) diagnosis of idiopathic PSP in accordance to the NINDS-SPSP International Criteria (Litvan et al., 1996), b) age between 55 and 85 c) ability to walk unassisted for at least 6 meters, d) stable dopaminergic drugs dosage in the month preceding the admission to the study. Exclusion criteria: a) any others significant neurological or orthopedic disorders, b) osteoarthritis, osteoporosis, cutaneous lesions and/or other pressure wounds, c) body weight exceeding 135 kg (the weight limit for the use of Lokomat®), respiratory and cardiovascular diseases.
  Interventions: Other: MIRT
- MIRT+Lokomat group (Experimental): This group underwent a 4-weeks MIRT involving the use of Lokomat® for 5 days per week in spite of treadmill-plus.
  Inclusion criteria: a) diagnosis of idiopathic PSP in accordance to the NINDS-SPSP International Criteria (Litvan et al., 1996), b) age between 55 and 85 c) ability to walk unassisted for at least 6 meters, d) stable dopaminergic drugs dosage in the month preceding the admission to the study. Exclusion criteria: a) any others significant neurological or orthopedic disorders, b) osteoarthritis, osteoporosis, cutaneous lesions and/or other pressure wounds, c) body weight exceeding 135 kg (the weight limit for the use of Lokomat®), respiratory and cardiovascular diseases.
  Interventions: Other: MIRT+Lokomat

INTERVENTIONS:
Other: MIRT — It consists of a 4-weeks physical therapy which entails four daily sessions for five days. All treatments are performed in aerobic condition. The duration of each session, including recovery periods, is about one hour. The first session consists of a one-to-one session with physical therapist. The second session includes aerobic and repetitive exercises to improve balance and gait using different devices: a posturographic platform with visual cues, cycloergometer, treadmill-plus. The third is a session of occupational therapy. The last session includes one hour of speech therapy.
  All patients undergo 20-minutes treadmill-plus training per day, 5 times a week, for 4 weeks.
  Arms: MIRT group
Other: MIRT+Lokomat — It consists of a 4-weeks physical therapy which entails four daily sessions for five days. All treatments are performed in aerobic condition. The duration of each session, including recovery periods, is about one hour. The first session consists of a one-to-one session with physical therapist. The second session includes aerobic and repetitive exercises to improve balance and gait using different devices: a posturographic platform with visual cues and cycloergometer. The third is a session of occupational therapy to improve autonomy in activities of daily life. The last session includes one hour of speech therapy. All patients undergo 20-minutes Lokomat® training per day in spite of treadmill-plus.
  Arms: MIRT+Lokomat group

SUMMARY:
The investigators evaluate whether an aerobic, intensive, goal based and multidisciplinary rehabilitation treatment, previously conceived for Parkinson's disease, is effective for patients with progressive supranuclear palsy and whether a driven gait orthosis (Lokomat) can provide further benefits.

ELIGIBILITY:
Inclusion Criteria:

a) diagnosis of PSP in accordance to the NINDS-SPSP International Criteria (Litvan et al., 1996), b) age between 55 and 85 c) ability to walk unassisted for at least 6 meters, d) stable dopaminergic drugs dosage in the month preceding the admission to the study

Exclusion Criteria:

a) any others significant neurological or orthopedic disorders, b) osteoarthritis, osteoporosis, cutaneous lesions and/or other pressure wounds, c) body weight exceeding 135 kg (the weight limit for the use of Lokomat®), respiratory and cardiovascular diseases.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
PSPRS | One month
  PSP Rating Scale

SECONDARY OUTCOMES:
BBS | One month
  Berg Balance Scale
NoF | One month
  Number of falls

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Frazzitta, MD, Principal Investigator — Ospedale generale di Zona "Moriggia-Pelascini", Gravedona ed Uniti 22015 - CO, Italy
Locations (1):
- Ospedale Generale di Zona "Moriggia-Pelascini", Gravedona, Como, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Clerici I, Ferrazzoli D, Maestri R, Bossio F, Zivi I, Canesi M, Pezzoli G, Frazzitta G. Rehabilitation in progressive supranuclear palsy: Effectiveness of two multidisciplinary treatments. PLoS One. 2017 Feb 3;12(2):e0170927. doi: 10.1371/journal.pone.0170927. eCollection 2017. PMID 28158197